CLINICAL TRIAL: NCT02603159
Title: Different Cycles of Capecitabine Usage in Esophageal Cancer Concurrent Chemoradiotherapy
Acronym: DCECRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Capecitabine and esophageal
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Stage III Esophageal Squamous Cell Carcinoma; Stage II Esophageal Squamous Cell Carcinoma
Keywords: Chemoradiotherapy; Esophageal Squamous Cancer; Capecitabine
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine-5 weeks-radiotherapy (Experimental): Capecitabine 5 weeks : 625mg/m2, bid d1-5; q1w, po,5 weeks in total, radiotherapy： 50Gy ，2 Gy/d，5d/w.
  Interventions: Drug: Capecitabine(Aibin); Radiation: radiotherapy
- Capecitabine-10 weeks-radiotherapy (Active Comparator): Capecitabine 10 weeks : 625mg/m2, bid d1-5; q1w, po,10 weeks in total, radiotherapy： 50Gy ，2 Gy/d，5d/w.
  Interventions: Drug: Capecitabine(Aibin); Radiation: radiotherapy

INTERVENTIONS:
Drug: Capecitabine(Aibin) — Capecitabine(Aibin)：625mg/m2, bid d1-5; q1w, po,5 or 10 weeks in total
  Other Names: Aibin
Radiation: radiotherapy — Concurrent radiotherapy： 50Gy in total，2 Gy/d，5d/w，Until disease progression or unacceptable toxicity
  Other Names: radiation therapy

SUMMARY:
Definitive chemoradiotherapy with cisplatin with cisplatin plus 5-fluorouracil is the standard in Western countries in esophagus cancer.But in China because of its toxic reaction, most of patients stop the halfway.Because low toxicity, Capecitabine is widely used in the chemotherapy of esophageal cancer.

The purpose of this experiment was to study the different cycle on capecitabine with chemotherapy for esophageal cancer chemoradiation effect.We are prepared to within 2 years study recruited 200 patients with esophageal cancer.The primary endpoint is overall survival and the secondary endpoints include progression-free survival, response rate,pathologic complete response rate and adverse events.

DETAILED DESCRIPTION:
We recruited the patients who were pathologically confirmed with esophageal squamous cell carcinoma from the Oct 2014. The the patients was divided into two groups. Group 1: Capecitabine + chemoradiation, radiation at the end of the stop using capecitabine. Group 2: Capecitabine + chemoradiation, at the end of the radiotherapy with capecitabine consolidating treatment for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age 45-75years old
* Histologically proven squamous cell carcinoma of the esophagus
* the tumor was in T2-4N0-2M0
* The patients have not received the surgery or chemo-radiotherapy.
* Hb≥80g/L, absolute neutrophil count ≥1.5×109/L, Plt≥90×109/L,
* ALT、AST≤2.5*N,Cr≤1.5*N.
* performance status score 0-2

Exclusion Criteria:

* pregnant, lactating women
* Oxaliplatin or fluorouracil Allergy or metabolic disorders
* Radiotherapy contraindications
* History of organ transplantation
* Brain metastasis
* The peripheral nervous system disorders
* Severe infection
* Oral capecitabine who have difficulty with,such as dysphagia,The activities of digestive ulcer, Gastrointestinal bleeding
* Severe chronic diseases, such as, hepatopathy, nephropathy, respiratory disease,high blood pressure, diabetes.
* Other malignant tumor in recent 5 years.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
overall survival, OS | 2 years

SECONDARY OUTCOMES:
progression-free survival | 2 years
overall remission rate, ORR | 16 weeks
serious adverse event | 16 weeks
quality of life, Qol | 16 weeks
pathologic complete response rate | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Science and Technology; Tanyou Shan, Master, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Xiaoshan Feng, Doctor, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Jiachun Sun, Doctor, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xinshuai Wang, Doctor, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Guoqiang Kong, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xiaozhi Yuan, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Ruinuo Jia, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Zhuo, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Jing Ren, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Ruina Yang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yali Zhang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yongxuan Liu, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Wei Wang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Wang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Weijiao Yin, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Shiyuan Song, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

REFERENCES:
- [Background] Park JW, Kim JH, Choi EK, Lee SW, Yoon SM, Song SY, Lee YS, Kim SB, Park SI, Ahn SD. Prognosis of esophageal cancer patients with pathologic complete response after preoperative concurrent chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):691-7. doi: 10.1016/j.ijrobp.2010.06.041. Epub 2010 Oct 1. PMID 20888705